CLINICAL TRIAL: NCT07184021
Title: Neoadjuvent Dose-dense Gemcitabine and Cisplatin In Muscle Invasive Bladder Cancer:Results of a Phase 2 Trial
Brief Title: Neoadjuvent Dose-dense Gemcitabine and Cisplatin In Muscle Invasive Bladder Cancer
Acronym: No Acronym
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal Ali Suliman, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Early Urinary bladder cancer
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Type of Study:
  Prospective, single-arm, interventional study evaluating the safety, feasibility, and pathological response of dose-dense neoadjuvant gemcitabine and cisplatin in muscle-invasive bladder cancer.
  2.4. 2- Study Setting: Clinical Oncology department, Assiut University Hospitals 2.4. 3- Study subjects:
  1. Inclusion criteria:
     * Histologically confirmed urothelial carcinoma of the bladder, clinical stage T2-T4a, N0-N1, M0.
     * Eligible and fit for cisplatin-based chemotherapy (e.g., creatinine clearance ≥ 60 mL/min).
     * Candidate for radical cystectomy after neoadjuvant treatment.
     * ECOG performance status 0-1.
     * Adequate bone marrow, liver, and renal function as per institutional standards.
  2. Exclusion criteria:
     * Histology predominantly other than urothelial carcinoma (e.g., small cell, squamous cell ≥50%).
     * Clinical or radiological evidence of distant metastases (M1).
     * Prior systemic chemotherapy or radiotherapy for bladder cancer.
     * Signific
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Dose-Dense Gemcitabine and Cisplatin (DDGC) (Experimental): Participants will receive four cycles of dose-dense gemcitabine and cisplatin (DDGC) prior to radical cystectomy. Each cycle consists of gemcitabine 1200 mg/m² intravenously on days 1 and 8, and fractionated cisplatin 35mg/m² intravenously on day 1and 8, repeated every 14 days. Pegfilgrastim 6 mg subcutaneously will be administered on day 2 of each cycle for growth factor support. Radical cystectomy will be performed 4-6 weeks after completion of chemotherapy.
  Interventions: Drug: Gemcitabine and Cisplatin (DD GC)

INTERVENTIONS:
Drug: Gemcitabine and Cisplatin (DD GC) — Participants will receive neoadjuvant ddGC, consisting of gemcitabine and cisplatin administered at shortened intervals (e.g., gemcitabine 1200 mg/m² on days 1 and 8, fractionated cisplatin 35 mg/m² on day 1and 8, every 14 days) with appropriate growth factor support. A total of four cycles are planned before radical cystectomy.

SUMMARY:
To evaluate the feasibility, safety, and pathological response of dose-dense neoadjuvant gemcitabine and cisplatin in patients with muscle-invasive bladder cancer, with the goal of improving tumor downstaging and optimizing outcomes before radical cystectomy.

DETAILED DESCRIPTION:
Muscle-invasive bladder cancer (MIBC) poses a significant therapeutic challenge due to its high risk of progression and metastasis. Radical cystectomy remains the cornerstone of curative treatment; however, many patients relapse due to undetected micrometastases at diagnosis. To address this, neoadjuvant chemotherapy (NAC) with cisplatin-based combinations has been established as standard care, demonstrating improved pathological downstaging and survival outcomes compared to surgery alone (Yin et al., 2020; Necchi et al., 2017).

Gemcitabine and cisplatin (GC) is widely favored in NAC because of its comparable efficacy to older regimens and a more favorable toxicity profile (Galsky et al., 2016). However, conventional schedules may be limited by treatment delays and incomplete cycles, often due to cumulative toxicities or patient frailty. Dose-dense chemotherapy-delivering the same drugs at shorter intervals with growth factor support-has been proposed to improve outcomes by intensifying dose intensity and reducing tumor repopulation between cycles (Zargar et al., 2018; Kulkarni et al., 2020).

Evaluating dose-dense GC in the neoadjuvant setting aims to balance efficacy and tolerability, potentially increasing rates of complete pathological response and improving long-term survival. This protocol seeks to explore the feasibility, safety, and oncological benefit of this approach in patients with MIBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed urothelial carcinoma of the bladder, clinical stage T2-T4a, N0-N1, M0.
* Eligible and fit for cisplatin-based chemotherapy (e.g., creatinine clearance ≥ 60 mL/min).
* Candidate for radical cystectomy after neoadjuvant treatment.
* ECOG performance status 0-1.
* Adequate bone marrow, liver, and renal function as per institutional standards.

Exclusion Criteria:

Histology predominantly other than urothelial carcinoma (e.g., small cell, squamous cell ≥50%).

* Clinical or radiological evidence of distant metastases (M1).
* Prior systemic chemotherapy or radiotherapy for bladder cancer.
* Significant renal impairm ent (creatinine clearance < 60 mL/min).
* ECOG performance status ≥ 2.
* Significant comorbidities contraindicating chemotherapy (e.g., uncontrolled cardiac disease, severe infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pT0N0) Rate | At the time of radical cystectomy (approximately 4-6 weeks after completion of neoadjuvant chemotherapy).
  Proportion of participants with no residual invasive or non-invasive tumor in the bladder and no lymph node involvement (ypT0N0) at the time of radical cystectomy, as determined by histopathological examination of the surgical specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Rayan, Professor, Study Director — Assiut University Hospitals, Faculty of medicine, Assiut University
Locations (1):
- Assiut university Hospital-Departement of clinical oncology., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Because of institutional policy and patient confidentiality considerations.

REFERENCES:
- See also: Assiut University Hospitals — https://www.aun.edu.eg/hospitals
- Available data/document: Study Protocol: Protocol draft available — https://www.aun.edu.eg/hospitals — Individual participant data and supporting documents will not be shared in order to protect patient confidentiality.